CLINICAL TRIAL: NCT04098484
Title: Biological Adaptations of Strength Training to Obese and Normal Weight Middle-aged Men
Brief Title: Biological Adaptations of Strength Training.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Athanasios Chatzinikolaou, Associate Professor, Democritus University of Thrace
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXERCISE-OBESITY-DUTH
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Obesity, training, inflammation, Liver, oxidative stress
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal-weight (Active Comparator): Subjects with a BMI of 18-25 kg/m2
  Interventions: Other: Control Trial; Other: Exercise Trial
- Obese (Experimental): Subjects with a BMI of > 30 kg/m2
  Interventions: Other: Control Trial; Other: Exercise Trial

INTERVENTIONS:
Other: Control Trial — Participants will abstain from exercise throughout a 3-month period
Other: Exercise Trial — Participants will execute a 3-month exercise training program

SUMMARY:
A two-trial repeated measures design will be employed in this investigation. Both the control trial and the exercise trial will last for 3 months. During a week before the start of the study, participants will complete dietary recalls and record their habitual physical activity using accelerometers. Thereafter, body composition, ultrasound imaging of the muscle and liver, biochemical and hematological markers were measured. This range of measurements will be repeated the ended each month for both trials. Control trial succeeds exercise trial. An exercise intervention program will take place in the second trial, three times a week.

DETAILED DESCRIPTION:
A sample size of 30 volunteers, aged 35-45 years, will participate in the present study. Of them, 15 will be normal weight and 15 will suffer from fatty liver disease (BMI 29-35 kg/m2, waist size >102 cm). The exclusion criteria will be a) medication, b) musculoskeletal problems that will prevent participation in the training program, c) known condition or medical condition preventing participation in the program e.g. hypertension, d) BMI> 35kg / m2, (e) a severe family medical history up to first degree relatives with cardiovascular disease and / or diabetes at the age of less than 65 for women and less than 55 years for men and (f) smoking. After informing and receiving a questionnaire and medical history, volunteers will sign for their participation in the survey.

A two-trial repeated measures design will be applied in this investigation. Both control and exercise trials will last for 3 months. During the week preceding the commencement of the study, participants will complete dietary recalls and will have their habitual physical activity monitored, by utilizing accelerometers. Thereafter, body composition, ultrasound imaging of muscle and liver, biochemical and hematological markers will be measured. The same measurements will be repeated at the end of each month, in both trials. Control trial will be executed prior to exercise trial. An exercise intervention program, combining strength and cardiovascular exercises performed three times a week, will take place in the exercise trial.

ELIGIBILITY:
Inclusion Criteria:

* no use of medication
* free of musculoskeletal limitations
* absence of a known condition or medical condition preventing participation in the program (e.g. hypertension)
* absence of a severe family medical history up to first degree relatives with cardiovascular disease and /or diabetes at the age of less than 65 for women and less than 55 years for men
* non-smokers

Exclusion Criteria:

* use of medication
* musculoskeletal limitations that will prevent participation in the training program
* known condition or medical condition preventing participation in the program (e.g. hypertension)
* a severe family medical history up to first degree relatives with cardiovascular disease and /or diabetes at the age of less than 65 for women and less than 55 years for men
* smoking

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-12-25 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in body composition | At baseline as well as at 1,5 and 3 months in both trials
  Body composition will be assessed using Dual-energy-X-ray Absorptiometry (DXA) instrumentation
Changes in HDL concentration | At baseline as well as at 1,5 and 3 months in both trials
  HDL concentration will be measured in blood
Changes in LDL concentration | At baseline as well as at 1,5 and 3 months in both trials
  LDL concentration will be measured in blood
Changes in total cholesterol | At baseline as well as at 1,5 and 3 months in both trials
  Total cholesterol levels will measured in blood
Changes in triglycerides | At baseline as well as at 1,5 and 3 months in both trials
  Triglycerides concentration will be measured in blood
Changes in free fatty acids | At baseline as well as at 1,5 and 3 months in both trials
  Free fatty acid concentration will be measured in blood
Changes in glucose | At baseline as well as at 1,5 and 3 months in both trials
  Glucose concentration will be measured in blood
Changes in glycosylated hemoglobin | At baseline as well as at 1,5 and 3 months in both trials
  Glycosylated hemoglobin levels will be measured in blood
Changes in insulin | At baseline as well as at 1,5 and 3 months in both trials
  Insulin concentration will be measured in blood
Changes in insulin resistance index | At baseline as well as at 1,5 and 3 months in both trials
  Insulin resistance index will be calculated through glucose and insulin values
Changes in White Blood Cells | At baseline as well as at 1,5 and 3 months in both trials
  White blood cells will be measured in bood samples
Changes in Red Blood Cells | At baseline as well as at 1,5 and 3 months in both trials
  Red blood cells will be measured in bood samples
Changes in Hemoglobin | At baseline as well as at 1,5 and 3 months in both trials
  Hemoglobin will be measured in blood samples
Changes in Hematocrit | At baseline as well as at 1,5 and 3 months in both trials
  Hematocrit levels will be measured in blood samples
Changes in transaminases | At baseline as well as at 1,5 and 3 months in both trials
  Transaminase levels will be measured in blood samples
Changes in C-reactive protein | At baseline as well as at 1,5 and 3 months in both trials
  C-reactive protein levels will be measured in blood samples
Changes in total antioxidant capacity | At baseline as well as at 1,5 and 3 months in both trials
  Total antioxidant capacity will be assessed in plasma
Changes in glutathione | At baseline as well as at 1,5 and 3 months in both trials
  Oxidized (GSH) and reduced (GSSG) glutathione will be measured in red blood cell lysate
Changes in protein carbonyls | At baseline as well as at 1,5 and 3 months in both trials
  Protein carbonyl formation will be measured in serum
Changes in thiobarbituric acid reactive substances (TBARS) | At baseline as well as at 1,5 and 3 months in both trials
  TBARS will be measured in serum
Changes in catalase | At baseline as well as at 1,5 and 3 months in both trials
  Catalase activity will be measured in serum
Changes in fatty infiltration of the liver | At baseline as well as at 1,5 and 3 months in both trials
  Fatty infiltration of the liver will be assessed by ultrasound imaging of liver
Changes in bone status | At baseline as well as at 1,5 and 3 months in both trials
  Bone mineral density and bone mineral content will be assessed in hole body, spine and hips using DXA

SECONDARY OUTCOMES:
Changes in body weight | At baseline as well as at 1,5 and 3 months in both trials
Changes in muscle architecture | At baseline as well as at 1,5 and 3 months in both trials
  Muscle architecture of quadriceps will be assessed by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Maria Protopapa, PhDc, Principal Investigator — Democritus University of Thrace, School of Physical Education and Sports Science
Locations (1):
- Democritus University of Thrace, School of Physical Education and Sports Science, Komotini, Greece